CLINICAL TRIAL: NCT06895473
Title: A Phase 2 Study of Prophylactic IT Chemotherapy to Prevent High-Grade Chimeric Antigen Receptor (CAR) T-Cell-Associated Neurotoxicity Syndrome
Brief Title: Intrathecal Cytarabine, Methotrexate, and Hydrocortisone for the Prevention of High-Grade Chimeric Antigen Receptor T-Cell-Associated Neurotoxicity Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Stephen Spurgeon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00028106; NCI-2025-00937 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00028106 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Specimen Handling; Cytarabine; Spinal Puncture; Methotrexate; merphos; Hydrocortisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive Care (cytarabine, methotrexate, hydrocortisone) (Experimental): Patients receive cytarabine IT, methotrexate IT, and hydrocortisone IT over 3-5 minutes via LP on day 4 post-SOC CAR T-cell therapy in the absence of unacceptable toxicity or development of ICANS. Patients who do not develop ICANS of any grade, also receive hydrocortisone IT on day 7 post SOC CAR T-cell therapy. Additionally, patients undergo CSF sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cytarabine; Procedure: Lumbar Puncture; Drug: Methotrexate; Drug: Therapeutic Hydrocortisone

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid

SUMMARY:
This phase II trial tests how well cytarabine (Ara-C), methotrexate, and hydrocortisone given between the spinal cord and the membranes that protect it (intrathecal [IT]) works in preventing high-grade immune effector-associated neurotoxicity syndrome (ICANS) in patients receiving chimeric antigen receptor (CAR) T-cell therapy. ICANS is a challenging complication of CAR T-cell therapy that causes neurological effects varying from mild headaches or temporary confusion to hallucinations, swelling in the brain, and seizures. Between 20%-70% of patients receiving CAR T-cell therapy show symptoms of neurotoxicity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of IT chemotherapy in the prevention of high grade ICANS.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of IT chemotherapy in the prevention of any grade ICANS.

II. To evaluate safety of IT chemotherapy. III. To evaluate the effect of IT chemotherapy on corticosteroid use. IV. To evaluate the effect of IT chemotherapy on anakinra use.

EXPLORATORY OBJECTIVES:

I. To evaluate the effect of IT chemotherapy on time to ICANS onset. II. To evaluate the effect of IT chemotherapy on duration of ICANS. III. To evaluate the burden of treatment mediated serious adverse events (SAEs).

OUTLINE:

Patients receive cytarabine IT, methotrexate IT, and hydrocortisone IT over 3-5 minutes via lumbar puncture (LP) on day 4 post-standard of care (SOC) Axi-cel (Yescarta) or Brexu-cel (Tecartus) in the absence of unacceptable toxicity or development of ICANS. Patients who do not develop ICANS of any grade, also receive hydrocortisone IT on day 7 post SOC CAR T-cell therapy. Additionally, patients undergo cerebrospinal fluid (CSF) sample collection throughout the study.

After completion of study treatment, patients are followed for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent. Participant or legally authorized representative (LAR) must provide written informed consent prior to any study-specific procedures or interventions
* Age ≥ 18 years. All genders, races, and ethnic groups will be included
* Must be receiving SOC Yescarta® or Tecartus® in the inpatient setting
* Agree to adhere to institutional guidelines for contraception during the first 30 days post CAR-T

  * Rationale for eligibility criteria based on contraception and pregnancy (both participants and partners of a sperm-producing participant): It shall be known to all participants that the effects of CAR-T or IT chemotherapy on the developing human fetus are unknown. For this reason, persons of reproductive potential must agree to use adequate contraception. Should a participant or participant's sexual partner become pregnant or suspect a pregnancy while participating in this study, the individual should inform their treating physician immediately
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Platelet count > 50,000/mm^3 (μL)
* Adequate coagulation tests including international normalized ratio (INR) < 1.6 and fibrinogen > 100

Exclusion Criteria:

* Active/concurrent diagnosis of any central nervous system (CNS) hematologic malignancy

  * History or presence of CNS disorder such as poorly controlled seizure disorder (seizure within the 12 months), transverse myelitis, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* Known history of hypersensitivity to IT chemotherapy
* Subject has a contraindication to LP including:

  * Presence of a posterior fossa mass
  * Skin infection near puncture site
  * Uncorrected bleeding diathesis
  * Suspicion of increased intracranial pressure
  * Acute spinal cord trauma
* Subject is receiving an antiplatelet and/or anticoagulant that cannot be held prior to LP according to best available evidence
* Known bleeding disorders
* Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgement, make the participant inappropriate for study participation or would put the participant at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of American Society for Transplantation and Cellular Therapy (ASTCT) ≥ grade 3 immune-effector cell associated neurotoxicity syndrome (ICANS) | From first dose of intrathecal (IT) chemotherapy (chimeric antigen receptor [CAR]-T day 4) to CAR-T day 30
  Will be reported using the efficacy set. Point estimate, along with exact two-sided 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Incidence of ASTCT any grade ICANS | From first dose of IT chemotherapy (CAR-T day 4) to CAR-T day 30
  Will be reported using the efficacy set. Point estimate, along with exact two-sided 95% confidence interval will be reported.
Incidence of lumbar puncture/IT treatment related adverse events (AEs) and serious adverse events (SAEs) | From first dose of IT chemotherapy (CAR-T day 4) to CAR-T day 30
  Will be reported using the safety set. AEs will be tabulated by the Medical Dictionary for Regulatory Activities version (v) 21.1. preferred term and system organ class and a preferred term. The severity of the AE will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version (CTCAE) v 5.0. Descriptive statistics using the safety evaluable population, will be used to report on all on-study AEs, grade 3-4 AEs, treatment-related AEs, grade 3-4 treatment-related AEs, SAEs, treatment-related SAEs, and AEs leading to discontinuation per CTCAE v 5.0. Grade 3-4 laboratory abnormalities will be summarized using worst grade NCI CTCAE v 5.0 criteria.
Mean (range) cumulative dose of corticosteroid use | From first dose of IT chemotherapy (CAR-T day 4) to CAR-T day 30
  Will be reported using the efficacy set. The cumulative dose will be calculated as the sum of all corticosteroid administered over the study period, expressed in milligrams (mg) of prednisone-equivalent.
Incidence of anakinra use | From first dose of IT chemotherapy (CAR-T day 4) to CAR-T day 30
  Will be reported using the efficacy set. Point estimate, along with exact two-sided 95% confidence interval will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States